CLINICAL TRIAL: NCT03905304
Title: A Prospective, Randomized, Multi-center, Phase III, Double-Blind, Activi Controlled, Parallel-group Study to Evaliate the Efficacy and Safety of MEDITOXIN® Comparison With BOTOX® in Treatment of Cervical Dystonia
Brief Title: Efficacy and Safety of MEDITOXIN® in Cervical Dystonia
Acronym: CD Phase III
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medy-Tox (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MT_PRT_CD01
Record Dates: First submitted 2019-03-27; First posted 2019-04-05 (Actual); Last update posted 2019-04-08 (Actual); Status verified 2019-04

CONDITIONS: Cervical Dystonia
Keywords: CD phase III
MeSH Terms: conditions — Torticollis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Meditoxin (Experimental): Meditoxin administered 200U~300U, single-dose administration.
  Interventions: Biological: Medytoxin
- Botox (Active Comparator): Botox administered 200-300U, single-dose administration.
  Interventions: Biological: Botox

INTERVENTIONS:
Biological: Medytoxin — Intramuscular injection up to 300U.
  Other Names: botulinum type A toxin
  Arms: Meditoxin
Biological: Botox — Intramuscular injection up to 300U.
  Other Names: botulinum type A toxin
  Arms: Botox

SUMMARY:
The purpose of this study is to test the hypothesis that the efficacy and safety of Meditoxin® are not inferior to Botox®'s in the treatment of Cervical Dystonia.

DETAILED DESCRIPTION:
The allocated subject is injected Investigational Product(Meditoxin® or Botox®) 200~300U in cervical muscles. The efficacy and safety are evaluated for 12weeks through 4 follow up visits.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged between 20 and 75.
* Patient who is diagnosed with primary cervical dystonia over 1 year.
* Patients whose total score is over 20 in TWSTRS and the severity score is over 10 in TWSTRS.
* For patients with prior treatments of Botox®, over 12 weeks have passed.
* Patients who voluntarily sign the informed consent
* Patients who can comply with the study procedures and visit schedule

Exclusion Criteria:

* Patient who has been diagnosed with pure anterocollis.
* Patient who has been diagnosed with neuromuscular disorder(myasthenia gravis, Eaton-Lambert syndrome, amyotrophic lateral sclerosis, etc.)\
* Severe respiratory function disorder or dysphasia
* Allergy in Investigational Product.
* Pregnant women, breast feeding women and patients disagreeing to use an acceptable contraception method
* Investigator's decision.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2013-01-09 (Actual); Primary Completion 2014-07-30 (Actual); Study Completion 2014-08-05 (Actual)

PRIMARY OUTCOMES:
Change in TWSTRS score | 1 month
  Change in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) total score after 1 month of administration. The scale consists scores from 0 to 35 which corresponds to disorder severity, 35 being the most severe.

SECONDARY OUTCOMES:
Safety Analysis of Investigational Product: Number of adverse events occuring during the clinical trial | 1, 2, 3 months
  Number of adverse events occuring during the clinical trial.
Change in TWSTRS score | 1, 2, 3 months
  Change in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) score after 1, 2, and 3 month of administration. The scale consists scores from 0 to 35 which corresponds to disorder severity, 35 being the most severe.